CLINICAL TRIAL: NCT05506111
Title: Erfassung Des Low Anterior Resection Syndroms Nach Rektumresektion Bei Patienten Mit Einem Rektumkarzinom - Eine österreichweite Multi-center Studie
Brief Title: Low Anterior Resection Syndrome After Rectum Resection for Rectal Carcinoma.
Acronym: LARS-Austria
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Paracelsus Medical University (Other)
Collaborators: Department of Surgery Hospital of St. John of God, Graz (Unknown); Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Jaroslav Presl, Principal Investigator, Paracelsus Medical University
Other Study IDs: 1110/2021
Record Dates: First submitted 2022-07-22; First posted 2022-08-18 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Low Anterior Resection Syndrome; Quality of Life; Incontinence
MeSH Terms: conditions — Low Anterior Resection Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The ACO-ASSO (Austrian Society of Surgical Oncology) colorectal group and Austrian Working Group for Coloproctology present the LARS Austria study. It is a prospective, multicenter observational study. The primary objective of this study is to collect information about LARS (LARS score) and QoL (EORTC -CR29) in patients with non-metastatic rectal cancer who received therapy. As a secondary objective, the impact of radiotherapy on the occurrence of LARS will be investigated.

DETAILED DESCRIPTION:
All consecutive patients with biopsy verified rectal cancer (≤16cm from anocutaneous line) can be included in the study. For the study, tumors whose aboral margin, when measured with a rigid rectoscope, is 16 cm or less from the anocutaneous line will be included. Thus, only histologically verified tumors of the lower (<6 cm), middle (6<12 cm) and upper (12-16cm) rectal thirds are included.

Patients will be included after the indication for further therapy has been established in the tumor board according to guideline criteria and after signing the participation consent. The collection of study relevant data will be performed according to the following scheme:

Group 1 = patients without neoadjuvant radiochemotherapy (RCHT). Collection of data and questionnaires before surgery and 3, 6, and 12 months after index surgery (if no protective stoma).

OR Collection of data and questionnaires before surgery and 3, 6, or 12 months after stoma re-operation (if protective stoma).

Group 2 = patients with neoadjuvant RCHT/ definitive RCHT=watch and wait. Collection of data and questionnaires before RCHT and before surgery or after RCHT and 3, 6, or 12 months after index surgery (if no protective stoma).

OR Collection of data and questionnaires before RCHT and before operation=surgery(OP) or after RCHT and 3, 6 or 12 months after stoma closure (if protective stoma) OR Collection of data and questionnaires before RCHT and 3, 6 and 12 months after RCHT (if no surgery)

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 99 years
* Patients with biopsy-verified rectal cancer.
* Patients scheduled for elective sphincter-preserving rectal surgery
* Patients scheduled for neoadjuvant RCTx (Chemo-radiation) (concept: short course radiation, conv.

fractionated RCTx, total neoadjuvant therapy(TNT))

* Signed consent (ICF)

Exclusion Criteria:

* Patients younger than 18 years
* Patients without signed informed consent
* Metastatic carcinoma
* terminal colostomy ( APR (abdominoperineal resection),...)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients with a bioptically verified rectal carcinoma ≤16 cm from anocutaneous line) can be included in the study. Patients will be included only after the indication for further therapy has been established in the tumor board according to guideline criteria and after signing the informed consent form.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-07-18 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Detection of Low Anterior Resection Syndrome (LARS) after anterior rectal resection. | 3 months after the rectum resection or after the closure of a protective ileostomy or after an Chemoradiation in case of watch and wait
  Occurrence of Low Anterior Resection Syndrome (LARS) will be measured with an LARS Score. The score ranges from 0 to 42 is divides into no LARS (0 to 20 points), minor LARS (21 to 29 points), and major LARS (30 to 42 points)
Detection of Low Anterior Resection Syndrome (LARS) after anterior rectal resection. | 6 months after the rectum resection or after the closure of a protective ileostomy or after an Chemoradiation in case of watch and wait
  Occurrence of Low Anterior Resection Syndrome (LARS) will be measured with an LARS Score. The score ranges from 0 to 42 is divides into no LARS (0 to 20 points), minor LARS (21 to 29 points), and major LARS (30 to 42 points)
Detection of Low Anterior Resection Syndrome (LARS) after anterior rectal resection. | 12 months after the rectum resection or after the closure of a protective ileostomy or after an Chemoradiation in case of watch and wait
  Occurrence of Low Anterior Resection Syndrome (LARS) will be measured with an LARS Score. The score ranges from 0 to 42 is divides into no LARS (0 to 20 points), minor LARS (21 to 29 points), and major LARS (30 to 42 points)

SECONDARY OUTCOMES:
Assessing the difference in LARS Score between the time of the diagnoses (baseline)and after the chemoradiation to identify the impact of the neoadjuvant Chemo-Radiation on LARS. | At the time of the diagnosis (baseline) and 6 to 8 weeks after an Chemo-Radiation, directly before the surgery respectively.
  Occurrence of Low Anterior Resection Syndrome (LARS) will be measured with an LARS Score. The score ranges from 0 to 42 is divides into no LARS (0 to 20 points), minor LARS (21 to 29 points), and major LARS (30 to 42 points)

OTHER OUTCOMES:
Recording the risk factors for the occurrence of LARS. | baseline
  Assessing the potential risk factors like patient age, tumour high, patient BMI, UICC Stage (Union Internationale Contre le Cancer).
Recording the risk factors for the occurrence of LARS. | up to 4 weeks after the intervention/surgery or at the time of discharge from the hospital (if hospital stay longer than 4 weeks)
  Assessing the potential risk factors like art of the operation, postoperative complications, protective stoma, chemo-radiation.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Riss, Prof. Dr., Study Chair — Medical University Wien, Department of Surgery; Felix Aigner, Prof. Dr., Study Director — Department of Surgery Hospital of St. John of God, Graz; Jaroslav Presl, Dr., Principal Investigator — Paracelsus Medical University Salzburg, Department of Surgery
Locations (3):
- Austria (3):
  - Department of Surgery Hospital of St. John of God, Graz, Graz
  - Department of Surgery, Paracelsus Medical University, Salzburg
  - Department of Surgery Medical University Vienna, Vienna